CLINICAL TRIAL: NCT03998553
Title: Study for Obtaining Mature Oocytes by in Vitro Maturation in Oocyte-donor Women
Acronym: IVM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1901-VLC-006-EB
Record Dates: First submitted 2019-06-03; First posted 2019-06-26 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Female Infertility
Keywords: OOCYTE ACTIVATION; IN VITRO MATURATION; OOCYTE RETRIEVAL; DONNOR; hMG-HP
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: Prospective and unicentric cohort pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: IN VITRO MATURATION AND OOCYTE ACTIVATION — This study aims to fine-tune the in vitro maturation (IVM) technique to achieve nuclear mature oocytes, i.e., to mature the oocytes up to the metaphase II stage. In addition, an artificial oocyte activation (AOA) will be carried out to check the cytoplasmic maturation of the oocytes, avoiding the generation of potentially viable embryos.

SUMMARY:
In vitro maturation (IVM) is a technique for obtaining potentially fertilizable oocytes from immature oocytes. An oocyte must be mature both nuclearly and cytoplasmically in order to be competent in the reproductive process. Nuclear maturation involves an oocyte in metaphase II stage and is easily evaluated for its morphology. However, cytoplasmic maturation can only be evaluated by in vitro fertilization of that oocyte A mature nuclear and cytoplasmic oocyte is one capable of producing a viable embryo. This study aims to fine-tune the in vitro maturation (IVM) technique to achieve nuclear mature oocytes, i.e., to mature the oocytes up to the metaphase II stage. In addition, an artificial oocyte activation (AOA) will be carried out to check the cytoplasmic maturation of the oocytes, avoiding the generation of potentially viable embryos.

The aim of this study is to evaluate the response to the strategy stimulation with highly purified human menopausal gonadotropin (hMG-HP) administered for three days, in association with a standard methodology of in vitro oocyte maturation (IVM), to be performed on oocyte donors.

The correct functioning of this IVM technique would mean a reduction in the costs of ovarian stimulation treatments, as lower doses and shorter stimulation times are required, which implies lower risks for women derived from the medication and less stress for them.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18-35 years who have belonged to the egg donation program.
* Donors who agree to participate in the pre-trial report and sign informed consent.
* Good previous documented response to ovarian stimulation (at least 10 oocytes total and/or 8 MII).
* Donors with at least one previous cycle of donation, in which all the oocytes obtained were fertilized in fresh
* Patients who come to their last cycle of donation allowed by law
* No personal or family medical disorders history.
* Body mass index between 18-28 kg/m2
* Normal uterus and ovaries, without organic pathology
* Non-polycystic-looking ovaries
* Antral follicle Count (AFC) > 12 from both ovaries on day 2-3 of the menstrual cycle.
* Normal Karyotype
* Negative values of infectious diseases (hepatitis B virus, hepatitis C virus, human immunodeficiency virus and syphilis)
* Analytical with CBC, hemostasis and biochemistry with parameters within normality

Exclusion Criteria:

* Any systemic or metabolic disorder that counterindicates the use of gonadotrophins.
* Any medical condition involving non-inclusion in the oocyte donation program
* Who are taking hormonal contraceptives in the last 3 months
* Severe male Factor (Semen < 3 million)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
rate of obtaining potentially competent oocytes | 6 months
  Number of potentially competent oocytes (after in vitro maturation and oocyte activation).

SECONDARY OUTCOMES:
Oocyte retrieval rate | 6 months
  Number of Oocyte retrieved per punctured follicle.
Artificial oocyte activation rate. | 6 months
  Number of activated oocyte obtained.
In vitro nuclear maturation rate. | 6 months
  Number of oocyted with matured nucleous.
Fertilization rate | 6 months
  Number of Fertilized oocytes obtained in a previous cycle of fresh donation of donor versus the obtained on in vitro maturation cycle.
Mature oocytes rate | 6 months
  Number of Mature oocytes obtained in of a previous cycle of fresh donation of donor versus the obtained on in vitro maturation cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- Ivi Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided